CLINICAL TRIAL: NCT01660906
Title: A Phase IV, Open-label, Multicenter Study of Dasatinib in Chronic-Phase Chronic Myeloid Leukemia (CP-CML) Patients With Chronic, Low-grade Non-Hematologic Toxicity to Imatinib
Brief Title: Phase IV, Open-label, Multicenter Study of Dasatinib in Chronic-Phase Chronic Myeloid Leukemia (CP-CML) Patients With Chronic, Low-grade Non-Hematologic Toxicity to Imatinib
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA180-400; 2011-006180-21 (EudraCT Number)
Record Dates: First submitted 2012-08-07; First posted 2012-08-09 (Estimated); Results first posted 2016-11-22 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Phase Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dasatinib (100 mg) (Experimental)
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib — tablets, oral, 100 mg, Once daily, Up to12 months on study,
  Other Names: Sprycel

SUMMARY:
This study proposes to evaluate the number of chronic, Grade 1 or 2, non-hematologic Adverse Events (AEs) that reduce in grade or resolve at 3 months after switching therapy from imatinib to dasatinib.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CML-CP patients achieving an optimal response to imatinib treatment with Grade 1 or 2 non-hematologic adverse events persisting for at least 2 months or recurring at least 3 times in the preceding 12 months, despite best supportive care
* Men and women with Chronic Myeloid Leukemia- Chronic Phase (CML-CP) Ph+ ≥ age 18
* Daily Eastern Co-Operative Group (ECOG) performance status = 0 - 2
* Patient willing and able to give informed consent
* Life expectancy > 6 months
* Adequate renal function
* Adequate hepatic function

Exclusion Criteria:

* Patients who are pregnant or breast feeding
* Men whose partner is unwilling to avoid pregnancy.
* Previous treatment with any other tyrosine-kinase inhibitor (TKI), except for imatinib
* Current grade 3 or 4 imatinib related adverse event
* Prior documented T315I mutation
* Prior diagnosis of accelerated phase or blast crisis CML
* Previous loss of complete hematologic response (CHR) or major cytogenetic response (MCyR) on imatinib
* Concurrent medical condition of uncontrolled infection, cardiovascular diseases of cardiac failure, congenital long QT syndrome, ventricular arrhythmias, prolonged QT interval, second or third degree heart block, uncontrolled angina, myocardial infarction (MI) in the last 6 months, uncontrolled hypertension, pulmonary arterial hypertension, pleural or pericardial effusions, or history of bleeding disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2012-12; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (21):
- United States (5):
  - Pacific Cancer Medical Center, Anaheim, California
  - Cancer Center Of Central Connecticut, Southington, Connecticut
  - St. Agnes Healthcare, Inc., Baltimore, Maryland
  - Promedica Hematology & Oncology Assoicates, Sylvania, Ohio
  - The University Of Texas Md Anderson Cancer Center, Houston, Texas
- France (5):
  - Local Institution, Créteil
  - Local Institution, Lille
  - Local Institution, Pierre-Bénite
  - Local Institution, Pringy
  - Local Institution, Vandœuvre-lès-Nancy
- Germany (5):
  - Local Institution, Cologne
  - Local Institution, Jena
  - Local Institution, Lübeck
  - Local Institution, Mannheim
  - Local Institution, Rostock
- Italy (5):
  - Local Institution, Catania
  - Local Institution, Florence
  - Local Institution, Napoli
  - Local Institution, Roma
  - Local Institution, Torino
- Local Institution, Seoul, South Korea

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 39 participants enrolled and were treated.
Groups:
- Dasatinib (100 mg): Dasatinib: A 100 mg tablet was taken orally once a day for up to 12 months while on study.
Period: Overall Study
Arm/Group | Dasatinib (100 mg)
Started | 39
Completed | 36
Not Completed | 3
Not completed — Discontinued due to study drug toxicity | 3

BASELINE CHARACTERISTICS:
Population: All treated participants.
Arm/Group | Dasatinib (100 mg)
Number analyzed (Participants) | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (15.13)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 27
  >= 65 years | 12
Gender [Count of Participants; unit: Participants]
  Female | 18
  Male | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 12
  Black or African American | 1
  American Indian or Alaska Native | 0
  Asian | 22
  Native Hawaiian or Other Pacific Islander | 0
  Other | 4
Median Time Since CML-CP Diagnosis [Median (Full Range); unit: months] — CML-CP, chronic myeloid leukemia-chronic phase
  months | 51.3 [3.9 to 214.6]
Median Duration of Imatinib Treatment [Median (Full Range); unit: months] | 51.2 [3.1 to 160.4]
Imatinib Dose at Baseline [Count of Participants; unit: Participants]
  < 400 milligrams | 19
  400 milligrams | 20
Best Baseline Response [Count of Participants; unit: Participants] — MR4.5, 4.5- log reduction in gene BCR-ABL transcript from the standardized baseline (0.0032% IS); MMR, Major Molecular Response = 3-log reduction in BCR-ABL gene transcripts from a standardized baseline; CCyR, complete cytogenetic response = criteria of 0% Philadelphia chromosome positive (Ph+) metaphases among cells in a bone marrow sample; PCyR, partial cytogenetic response = criteria of 1-35% Ph+ metaphases among cells in a bone marrow sample.
  3 patients did not have cytogenetic testing performed at screening and thus baseline responses could not be classified to a response category
  Participants
    MR4.5 | 10
    MMR | 20
    CCyR | 4
    PCyR | 2
    Cytogenetic Test Not Performed | 3

OUTCOME MEASURES:

1. Primary Outcome: The Number of Imatinib-related Adverse Events (AEs) That Were Resolved, Improved, Remained Unchanged, or Worsened After 3 Months of Dasatinib Treatment
Description: Dasatinib treatment was administered and its impact on the imatinib-related Grade 1/2 adverse events was assessed. The severity of an adverse event is ranked based on grades that range from 1 to 4. Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe, Grade 4= Potentially Life-threatening or disabling. Resolved, AE no longer present or resolution of imatinib-related chronic Grade 1 or Grade 2 non-hematologic AEs. Improved, AE grade reduced from Grade 2 to Grade 1. Unchanged, AE did not improve or worsen or no change in grade. Worsened, grade Increased.
Time Frame: 3 months after switch to dasatinib
Population: All treated participants.
Measure: Number; unit: adverse event(s)
Arm/Group | Dasatinib (100 mg)
Number analyzed (Participants) | 39
adverse event(s)
  Resolved | 91
  Improved | 2
  Unchanged | 27
  Worsened | 1

2. Secondary Outcome: Mean Change From Baseline in Patient Reported CML Symptom Severity and Interference by MD Anderson Symptom Inventory - Chronic Myeloid Leukemia (MDASI-CML) Score After Switching to Dasatinib
Description: The MD Anderson Symptom Inventory Chronic Myeloid Leukemia (MDASI-CML) is a validated questionnaire completed by study participants to assess symptom severity and symptom interference on daily function. These categories are divided into 5 domain summary scores: Core Symptom Severity Score, Interference Score, Symptom Severity Score, CML-Specific Symptom Severity Score, and 5 Most Severe Symptom Score. Scores were evaluated at baseline and after switching to Dasatinib on a range from 1 to 10; 1=not present/did not interfere, 10=as bad as you can imagine/interfered completely.
Time Frame: Baseline to 3, 6, 12 months
Population: All treated participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dasatinib (100 mg)
Number analyzed (Participants) | 39
units on a scale
  Core Symptom Severity Score, Month 3; n=37 | -1.35 (1.78)
  Core Symptom Severity Score, Month 6; n=36 | -1.44 (1.84)
  Core Symptom Severity Score, Month 12; n=37 | -1.06 (1.87)
  Interference Score, Month 3; n=37 | -1.24 (2.36)
  Interference Score, Month 6; n=35 | -1.28 (2.45)
  Interference Score, Month 12; n=36 | -1.30 (2.56)
  Symptom Severity Score, Month 3; n=37 | -1.73 (1.80)
  Symptom Severity Score, Month 6; n=36 | -1.80 (1.85)
  Symptom Severity Score, Month 12; n=37 | -1.46 (1.75)
  CML-specific Symptom Severity Score, Month 3; n=37 | -2.52 (2.35)
  CML-specific Symptom Severity Score, Month 6; n=36 | -2.60 (2.15)
  CML-specific Symptom Severity Score,Month 12; n=36 | -2.24 (1.87)
  5 Most Severe Symptom Score, Month 3; n=37 | -1.61 (1.76)
  5 Most Severe Symptom Score, Month 6; n=36 | -1.69 (1.84)
  5 Most Severe Symptom Score, Month 12; n=37 | -1.43 (1.72)

3. Secondary Outcome: Mean Change From Baseline in Patient Reported Quality of Life Measurements by The European Organization for Research and Treatment of Cancer - Quality of Life (QoL) Questionnaire (EORTC QLQ) Score After Switching to Dasatinib
Description: The EORTC QLQ-C30 questionnaire is completed by study participants to assess quality of life through nine multi-item scales: five functional scales (physical, role, cognitive, emotional and social functioning); three symptom scales (fatigue, pain and nausea/vomiting); and a global health status/QoL scale. Six single-item scales are also included (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). All of the scales and single-item measures were evaluated at baseline and after switching to Dasatinib as an average raw score that was standardized by transformation, so that final scores were on a range in score from 0 to 100. A high score for a functional scale represents a healthy level of functioning, a high score for the global health status/QoL represents a high QoL, but a high score for a symptom scale and single-item measures represents a high level of problematic symptomatology.
Time Frame: Baseline to 6, 12 months
Population: All treated participants
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dasatinib (100 mg)
Number analyzed (Participants) | 39
units on a scale
  Global Health Status/QOL, Month 6; n=36 | 0.46 (23.733)
  Global Health Status/QOL, Month 12; n=35 | 2.86 (27.782)
  Cognitive Functioning, Month 6; n=35 | 1.90 (20.119)
  Cognitive Functioning, Month 12; n=35 | 1.43 (18.245)
  Emotional Functioning, Month 6; n=35 | 11.19 (23.216)
  Emotional Functioning, Month 12; n=35 | 12.62 (25.595)
  Physical Functioning, Month 6; n=36 | -1.67 (20.923)
  Physical Functioning, Month 12; n=36 | 0.74 (19.241)
  Role Functioning, Month 6; n=36 | -4.17 (27.422)
  Role Functioning, Month 12; n=36 | 2.78 (23.401)
  Social Functioning, Month 6; n=35 | 13.81 (26.036)
  Social Functioning, Month 12; n=35 | 14.76 (24.512)
  Fatigue, Month 6; n=36 | -6.79 (20.102)
  Fatigue, Month 12; n=36 | -8.33 (21.639)
  Nausea and Vomiting, Month 6; n=36 | -9.72 (31.966)
  Nausea and Vomiting, Month 12; n=36 | -4.63 (30.760)
  Pain, Month 6; n=36 | -2.78 (38.318)
  Pain, Month 12; n=36 | -8.80 (25.350)
  Appetite Loss, Month 6; n=35 | 1.90 (29.085)
  Appetite Loss, Month 12; n=36 | 1.85 (29.755)
  Constipation, Month 6; n=36 | -0.93 (28.156)
  Constipation, Month 12; n=35 | 8.57 (23.351)
  Diarrhoea, Month 6; n=36 | 0.00 (36.515)
  Diarrhoea, Month 12; n=35 | -2.86 (40.722)
  Dyspnoea, Month 6; n=36 | 5.56 (36.947)
  Dyspnoea, Month 12; n=36 | 9.26 (39.530)
  Financial Difficulties, Month 6; n=35 | -10.48 (21.038)
  Financial Difficulties, Month 12; n=35 | -13.33 (18.436)
  Insomnia, Month 6; n=36 | 0.93 (42.528)
  Insomnia, Month 12; n=36 | -1.85 (38.991)

4. Secondary Outcome: Number of Participants With at Least 1 AE, Discontinuations Due to AE, Treatment-related AE, Serious Adverse Event (SAE), Treatment-related SAE, or Death as Outcome
Description: SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. Treatment-related=having certain, probable, possible, or missing relationship to study drug, dasatinib.
Time Frame: Date of first dose to 30 post last dose of study drug, an average of 3 years
Population: All treated participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Dasatinib (100 mg)
Number analyzed (Participants) | 39
Participants
  At least 1 AE | 37
  Discontinuation due to AE | 3
  Treatment-related AEs | 34
  SAEs | 11
  Treatment-related SAEs | 3
  Death | 0

5. Secondary Outcome: The Percentage of Participants With at Least 1 Imatinib-related Grade 1 or Grade 2 Chronic Adverse Events (AEs) That Improved Without Worsening Within 3 Months of Switching to Dasatinib
Description: Dasatinib treatment was administered and its impact on the Imatinib-related Grade 1/2 adverse events was assessed. The percentage of participants is based on the number that had pre-existing Imatinib-related AEs. Measure assesses the participants with reduction or improvement of at least 1 Imatinib-related Grade 1 or Grade 2 chronic AE, without a worsening of any Imatinib-related, chronic adverse events after Dasatinib treatment. The severity of an adverse event is ranked based on grades that range from 1 to 4. Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe, Grade 4= Potentially Life-threatening or disabling. Improved, AE grade reduced from Grade 2 to Grade 1. Worsened, Grade Increased. Confidence interval from Clopper-Pearson method.
Time Frame: 3 months
Population: All treated participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dasatinib (100 mg)
Number analyzed (Participants) | 39
percentage of participants | 87.1 [72.5 to 95.7]

6. Other Pre Specified Outcome: Number of Participants With a Major Molecular Response (MMR) and MR 4.5 After Switching to Dasatinib
Description: Molecular responses were assessed at 6 and 12 months after switching to dasatinib to determine if these baseline responses could be maintained. MR4.5, the number of treated participants with BCR-ABL transcripts ≤ 0.0032% (IS) at 6 and 12 months from the date of dasatinib initiation; MMR, Major Molecular Response = 3-log reduction in BCR-ABL gene transcripts from a standardized baseline.
Time Frame: 6 and 12 months
Population: All treated participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Dasatinib (100 mg)
Number analyzed (Participants) | 39
Participants
  MMR, Month 6 | 13
  MMR, Month 12 | 13
  MR4.5, Month 6 | 18
  MR4.5, Month 12 | 22

ADVERSE EVENTS:
Time Frame: Date of fist dose of study drug to 30 days post discontinuation of the last dose, an average of 3 years
Description: Study initiated: December 2012; Study Completion: October 2015
Groups:
- Dasatinib: Dasatinib: A 100 mg tablet was taken orally once a day for up to 12 months while on study.
Arm/Group | Dasatinib
Serious Adverse Events (participants affected / at risk) | 11/39
Other Adverse Events (participants affected / at risk) | 36/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib (N=39)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Haemorrhoids (Gastrointestinal disorders) | 2
Pneumonia (Infections and infestations) | 2
Appendicitis (Infections and infestations) | 1
Anal fissure (Gastrointestinal disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2
Rib fracture (Injury, poisoning and procedural complications) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Pyrexia (General disorders) | 1
Upper respiratory tract infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib (N=39)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2
Left ventricular hypertrophy (Cardiac disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 10
Anaemia (Blood and lymphatic system disorders) | 5
Asthenia (General disorders) | 2
General physical health deterioration (General disorders) | 2
Headache (Nervous system disorders) | 15
Blood urea increased (Investigations) | 2
Dizziness (Nervous system disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Nausea (Gastrointestinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10
Tendonitis (Musculoskeletal and connective tissue disorders) | 2
Blood creatinine increased (Investigations) | 3
Fatigue (General disorders) | 10
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Alanine aminotransferase increased (Investigations) | 2
Bronchitis (Infections and infestations) | 3
Depression (Psychiatric disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Hyperuricaemia (Metabolism and nutrition disorders) | 3
Paraesthesia (Nervous system disorders) | 3
Pericardial effusion (Cardiac disorders) | 3
Constipation (Gastrointestinal disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 11
Face oedema (General disorders) | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2
Pyrexia (General disorders) | 6
Rash (Skin and subcutaneous tissue disorders) | 10
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.